CLINICAL TRIAL: NCT01114048
Title: Early Response-adapted Intensification of Induction Chemotherapy in Patients With Newly Diagnosed Multiple Myeloma (MM) Who Are Eligible for Autologous Stem Cell Transplantation: Multicenter Phase 2 Study
Brief Title: Early Response-adapted Intensification of Induction Chemotherapy in Patients With Newly Diagnosed Multiple Myeloma (MM)
Acronym: KMM-97
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Je-Jung Lee, associate professor, Chonnam National University Hwasun Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMM-97
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Myeloma
Keywords: age under 65; Previous untreated
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Cyclophosphamide; Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Thalidomide, cyclophosphamide, dexamethasone, bortezomib — 1. Induction therapy with CTD regimen for 4 cycles Thalidomide 50-100 mg P.O. HS D 1~28 Cyclophosphamide 150 mg/m² P.O. D 1~4 Dexamethasone 20 mg/ m² IV or P.O. D 1~4, 15-18 Repeated every 28 days
  2. Intensification with Vel-CD regimen for 4 cycles (patients who fail to achieve more than PR after 2 cycles of CTD) Velcade 1.3 mg/m2 IV D1, 4, 8, 11 Cyclophosphamide 150 mg/m² P.O. D 1~4 Dexamethasone 20 mg/ m² IV or P.O. D1, 4, 8, 11 Repeated every 21 days
     * Bactrim prophylaxis during dexamethasone administration Acyclovir prophylaxis during velcade administration Aspirin medication during thalidomide administration

SUMMARY:
In this study, the investigators will analyze the long-term outcomes of remission and survival, and identify those with primary resistant disease as more likely to benefit from CTD (thalidomide, cyclophosphamide, dexamethasone) and early intensification of Vel-CD (bortezomib and CD) as induction chemotherapy followed by autologous stem cell transplantation for the patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
This study aims to assess the efficacy and toxicities of CTD and Vel-CD induction followed by high-dose therapy with autologous stem cell transplantation as a first line treatment for the patients with multiple myeloma.The investigators already investigated the thalidomide-based chemotherapy in patients with newly diagnosed MM. The combined regimen consisted of cyclophosphamide, thalidomide and dexamethasone (CTD) for induction treatment. CTD chemotherapy resulted in a favorable response with 79.4% overall response rate including 42.6% complete response (CR) or very good partial complete response (VGPR), and tolerable toxicity in MM patients. Moreover, CTD chemotherapy did not affect the yield of the stem cell collection.The investigators also published that the clinical efficacy and safety of a four-drug combination of bortezomib, cyclophosphamide, thalidomide, and dexamethasone was assessed for patients with relapsed or refractory multiple myeloma Vel-CTD chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed MM
2. Aged between 18 and 65 years old
3. With following measurable lesions (serum M-protein ≥ 1 g/dL or urine M-protein ≥ 400 mg/day, or free light chain ≥ 100 mg/L)

Exclusion Criteria:

1. Smoldering or indolent myeloma
2. ECOG performance status > 3 point
3. Known hypersensitivity to cyclophosphamide, thalidomide or dexamethasone
4. Peripheral neuropathy or neuropathic pain Grade 2 or higher as defined by NCI CTCAE version 3
5. Uncontrolled or severe cardiovascular disease, including MI within 6 months of enrolment, NYHA Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis, cardiac ejection fraction <0.5 : Severe conduction disorder : Hypotension (sitting systolic BP ≤ 100 mmHg and/or sitting diastolic BP ≤ 60 mmHg
6. Impaired hepatic function (AST or ALT ≥ x 3 upper normal, T-bilirubin ≥ x 2 upper normal)
7. Creatinine clearance < 20 ml/min
8. Corrected serum calcium ≥ 14 mg/dL
9. Sepsis or current active infection
10. Pregnancy or breast feeding
11. Uncontrolled Diabetes Mellitus
12. Previous history of Recurrent DVT or pulmonary embolism
13. Active ulcers detected by gastroscopy
14. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
15. Receipt of extensive radiation therapy within 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
response rate for induction chemotherapy | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do, South Korea